CLINICAL TRIAL: NCT00636896
Title: A Comparison of the Effects of Modafinil on Olanzapine Associated Eating Behaviors in Normal Human Subjects
Brief Title: Effects of Modafinil on Olanzapine Weight Gain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neuropsychiatric Research Institute, Fargo, North Dakota (Other)
Collaborators: Eli Lilly and Company (Industry); University of North Dakota (Other)
Responsible Party: James L. Roerig Pharm.D. Principal Investigator, University of North Dakota
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FID-US-X297
Record Dates: First submitted 2008-03-10; First posted 2008-03-17 (Estimated); Last update posted 2008-03-17 (Estimated); Status verified 2008-03

CONDITIONS: Weight Gain
Keywords: weight gain; olanzapine; atypical antipsychotic
MeSH Terms: conditions — Weight Gain | interventions — Olanzapine; Modafinil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Olanzapine 10 mg plus modafinil 200 mg
  Interventions: Drug: Olanzapine plus modafinil
- 2 (Placebo Comparator): Olanzapine plus Placebo
  Interventions: Drug: Olanzapine plus placebo

INTERVENTIONS:
Drug: Olanzapine plus modafinil — Olanzapine 10 mg/d plus modafinil 200 mg/d
  Other Names: Zyprexa; Provigil
  Arms: 1
Drug: Olanzapine plus placebo — Olanzapine 10 mg/d plus placebo
  Other Names: Zyprexa; Provigil
  Arms: 2

SUMMARY:
This study is designed as a 3 week, randomized, double blind, placebo controlled, trial. Olanzapine and modafinil will be titrated to 10mg and 200mg respectively. Feeding lab assessments will be conducted at baseline and endpoint. Assessments of hunger/satiety, kilocalories consumed and weight will be obtained. Plasma ghrelin and PYY3-36 levels will be drawn at baseline and endpoint prior to breakfast and two hours post.

Study hypothesis: The modafinil/olanzapine group will gain less weight than the olanzapine/placebo group over three weeks of drug intake.

DETAILED DESCRIPTION:
Atypical antipsychotics have become the drugs of choice in the treatment of schizophrenia as well as acute and maintenance therapy for bipolar disorder. In addition, affective disorders have been found to benefit from these agents (Masan 2004). These disorders represent chronic conditions that require extended treatment for years if not lifetimes. In light of the ever widening use of the atypicals, attention must now be focused on adverse reactions that may limit compliance with these agents. Weight gain and sedation have proven to be associated with many atypicals (Allison et al. 1999; Wirshing et al. 1999) including clozapine, olanzapine, risperidone and quetiapine. These side effects can reduce compliance and have detrimental effects on patient's health over long term treatment.

In our previous study, olanzapine and risperidone were demonstrated to affect eating behaviors and weight/BMI compared to placebo in a 2 week paradigm in normal healthy human subjects. Behaviors affected included appetite, reported calories consumed per day, and observed calories consumed in a feeding laboratory. No effects were seen on resting energy expenditure corrected for lean body weight. Also, sedation was reported in 81.3 and 75 % of the olanzapine and risperidone groups respectively. Sedation was the primary reason, in both groups, for medication dose reductions.

Weight gain and sedation have been postulated to be associated with the blockade of central nervous system (CNS) histamine-1 receptors (H1) by the atypical agents (Heisler 1998; Wirshing et al. 1999). In light of this postulated mechanism, it is reasonable to assume that overcoming the H1 blockade with a histamine agonist may aid in reducing these side effects to a tolerable level. Thus, the following study is proposed.

This study is designed as a randomized double blind, parallel group trial to evaluate the effect of modafinil (a proposed H1 agonist) vs. placebo on eating parameters, weight/BMI and sedation in healthy human subjects receiving olanzapine over a three week study period. This project utilizes the current state of the art feeding lab procedures, as reviewed by Mitchell and colleagues (Mitchell et al. 1998), to better characterize the effect of modafinil on olanzapine associated eating behavior. This project will help to determine the efficacy of utilizing a H1 agonist as an adjunctive medication in patients receiving atypical antipsychotic therapy to prevent weight gain and excess sedation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between the ages of 18 and 60 years.
* Women of child bearing potential must be practicing an accepted method of birth control (barrier method or oral contraceptive) and have a negative pregnancy test at baseline.
* Subjects must be of good general health by history and physical exam.

Exclusion Criteria:

* Subjects who are allergic to olanzapine or modafinil.
* Subjects with a history of a neuroleptic malignant syndrome.
* Subjects who have a body mass index at visit 2 less than 20 kg/m2 or greater than 27 kg/m2.
* Subjects who are restrictive eaters according to the restraint subscale of the Eating Disorder Evaluation (EDE).
* Women who are pregnant or nursing at the time of the study.
* Subjects who are lactose intolerant.
* Subjects with diabetes mellitus.
* Subjects experiencing clinically significant, unstable neurological, cardiac (including cardiac conduction defects), hepatic, renal disease or narrow angle glaucoma.
* Subjects diagnosed with anorexia nervosa, bulimia nervosa, or binge eating disorder.
* Subjects currently or with a past history of meeting DSM-IV diagnostic criteria for schizophrenia, schizoaffective disorder, bipolar disorder or substance abuse.
* Subjects who have participated in an investigational drug study in past 30 days.
* Subjects who are receiving any prescription medications other than oral contraceptives that would interact with the study medication or influence appetite or weight.
* Subjects who smoke or use any nicotine products.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2006-07; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Change in weight | 3 weeks

SECONDARY OUTCOMES:
Change in Kilocalories consumed | Over 3 weeks
Change in Epworth sleep scale | 3 weeks
Change in Food Craving Inventory | 3 weeks
Change in delta ghrelin | 3 weeks
Change in delta PYY3-36 | 3 weeks
Change in satiety ratings | 3 weeks
Change in hunger ratings | 3 weeks
Adverse effect comparison | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: James L Roerig, PharmD, Principal Investigator — University of North Dakota
Locations (1):
- Neuropsychiatric Research Institute, Fargo, North Dakota, United States

REFERENCES:
- [Background] Roerig JL, Steffen KJ, Mitchell JE, Crosby RD, Gosnell BA. A comparison of the effects of olanzapine and risperidone versus placebo on ghrelin plasma levels. J Clin Psychopharmacol. 2008 Feb;28(1):21-6. doi: 10.1097/jcp.0b013e3181613325. PMID 18204336
- [Background] Roerig JL, Mitchell JE, de Zwaan M, Crosby RD, Gosnell BA, Steffen KJ, Wonderlich SA. A comparison of the effects of olanzapine and risperidone versus placebo on eating behaviors. J Clin Psychopharmacol. 2005 Oct;25(5):413-8. doi: 10.1097/01.jcp.0000177549.36585.29. PMID 16160615
- See also: Neuropsychiatric Research Institute web page — http://www.nrifargo.com/